CLINICAL TRIAL: NCT03949010
Title: Investigation of the Effectiveness of Muscle Inhibition and Space Correction Techniques of Kinesiotaping Method in Female Patients With Myofascial Pain Syndrome Related to Upper Trapezius Active Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilşad Sindel (Other)
Responsible Party: Sponsor-Investigator, Dilşad Sindel, Professor, MD, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSCT&KMIT
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Female Patients With Myofascial Pain Syndrome (MPS) Related to Upper Trapezius Active Trigger Points (TP)
Keywords: Myofascial pain syndrome, kinesiotaping, upper trapezius, home exercise program
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping with space correction technique (Experimental)
  Interventions: Other: Kinesiotaping with space correction technique; Other: Home exercise program
- Kinesiotaping with muscle inhibition technique (Experimental)
  Interventions: Other: Kinesiotaping with muscle inhibition technique; Other: Home exercise program
- Home exercise program (Active Comparator)
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Kinesiotaping with space correction technique — Kinesiotaping with space correction technique twice per week for two weeks along with home exercise program
  Arms: Kinesiotaping with space correction technique
Other: Kinesiotaping with muscle inhibition technique — Kinesiotaping with muscle inhibition technique twice per week for two weeks along with home exercise program
  Arms: Kinesiotaping with muscle inhibition technique
Other: Home exercise program — Home exercise program which consists of stretching exercises towards neck area

SUMMARY:
To investigate the effectiveness of muscle inhibition and space correction techniques of kinesiotaping (KT) method; on pain, functional status and quality of life in female patients with myofascial pain syndrome (MPS) related to upper trapezius active trigger points (TP) in comparison to control group and to determine the advantage of each technique over another.

DETAILED DESCRIPTION:
The investigators conducted a prospective, randomized, controlled trial involving 93 female patients with MPS related to upper trapezius TPs and randomized the patients to KT treatment group with space correction technique and home exercise program (KSCT, n=20), KT treatment group with muscle inhibition technique and home exercise program (KMIT, n=24) and control group (CG, n=27) which received home exercise program only. Patients were evaluated by numerical rating scale (NRS) for their average and maximum pain intensity, Turkish version of neck disability index (NDI), and short form-36 (SF-36) scales. Statistical tests were conducted at the 0.05 significance level for all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* being female
* being aged between 18 and 45 years old
* not being in menopausal period
* having pain in upper trapezius region
* determining a taut band in examination
* having at least one active TP in this taut band
* the pain produced by palpation of this TP is the pain that the patient complains
* painfull restriction of cervical lateral flexion
* having pain score 4 or more according to NRS
* signing informed consent.

Exclusion Criteria:

* having major surgery or trauma related to the musculoskeletal system (primarily including the spine and upper extremity)
* having any operative history including the head and neck region
* having a neuromuscular disease
* having an active rheumatic disease
* having a systemic disease (diabetes, hypothyroidism, infection, malignancy...)
* having any pathology related to musculoskeletal diseases -especially including the cervical region- (cervical discopathy, cervical spondylosis, pathologies related to shoulder joint and surrounding soft tissues, scoliosis, kyphosis, limb length discrepancy, polio sequelae, developmental hip dysplasia...)
* having serious psychological problems (having score of 30 or more from Beck Depression Inventory)
* being obese (Body Mass Index≥30 kg/m2)
* having allergy to kinesiotapes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in pain related to myofascial pain syndrome due to upper trapezius active trigger points from baseline to first, second and six weeks | Initial assessment, First week, second week, sixth week
  Pain intensity mesaurement via Numerical Rating Scale, range between 0 to 10, higher scores indicating more pain intensity
Change in disability related to myofascial pain syndrome due to upper trapezius active trigger points from baseline to second and six weeks | Initial assessment, second week, sixth week
  Functional status measurement via Neck Disability Index
Change in quality of life affected by myofascial pain syndrome due to upper trapezius active trigger points from baseline to second and six weeks | Initial assessment, second week, sixth week
  Quality of life measurement via Short Form-36

IPD SHARING:
Plan to Share IPD: No